CLINICAL TRIAL: NCT06623396
Title: A Phase I Trial of Intraperitoneal Mesothelin-Targeted CAR T-Cell Therapy in Patients With Mesothelin-Positive Esophagogastric Adenocarcinoma With Peritoneal Carcinomatosis
Brief Title: A Study of Mesothelin-Targeted CAR T-Cell Therapy in People With Esophagogastric Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-214
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Mesothelin Positive; Mesothelin-Expressing Tumors; Esophageal Adenocarcinoma; Esophageal Adenocarcinomas; Esophagogastric Adenocarcinoma; Peritoneal Carcinomatosis; Breast Neoplasms; Diabetes Mellitus
Keywords: mesothelin positive; mesothelin-expressing tumors; esophageal adenocarcinoma; esophageal adenocarcinomas; esophagastric adenocarcinoma; peritoneal carcinomatosis; CAR T-Cell Therapy; 24-214
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Peritoneal Neoplasms; Breast Neoplasms; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with Mesothelin-Positive Esophagogastric Adenocarcinoma with Peritoneal Carcinomatosis (Experimental): Participants will be diagnoses with Mesothelin-Positive Esophagogastric Adenocarcinoma with Peritoneal Carcinomatosis
  Interventions: Biological: M28z1XXPD1DNR CAR

INTERVENTIONS:
Biological: M28z1XXPD1DNR CAR — Participants with esophagastric adenocarcinoma will be treated with an intraperitoneal infusion of different doses of autologous T cells that have been genetically modified ex vivo to express the M28z1XXPD1DNR CAR. The CAR T cells will be manufactured in MSK's Center for Cell Engineering.

SUMMARY:
Participants will have a sample of their white blood cells, called T cells, collected using a procedure called leukapheresis. The collected T cells will be sent to a laboratory at Memorial Sloan Kettering to be changed (modified) to become MSLN-targeted CAR T cells, the CAR T-cell therapy that participants will receive during the study. Participant study therapy will take about 3-4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* Diagnosis of pathologically confirmed EG adenocarcinoma
* Diagnosis of metastatic or recurrent disease
* ECOG performance status of 0-1
* Life expectancy of ≥4 months

Inclusion Criteria for Leukapheresis:

* Written informed consent for the study (from participant)
* Life expectancy of ≥4 months
* ECOG performance status of 0-1
* Histologic diagnosis that & >25% of the tumor expresses MSLN by IHC analysis. Archival tissue obtained up to 2 years before study enrollment is acceptable. IHC testing of a cell block from cytology (e.g., ascitic fluid) is acceptable if approved by the study pathologist. If adequate archival tissue is not available at screening, a fresh tumor biopsy should be obtained
* Stage IV disease with gross peritoneal carcinomatosis on imaging and/or microscopic peritoneal involvement by cytology or noted during diagnostic laparoscopy
* Disease progression or treatment intolerance after receiving at least 1 treatment regimen in the metastatic setting; patients with disease recurrence within 6 months of completing curative systemic therapy (chemotherapy, chemoradiation or adjuvant immunotherapy) are also eligible
* Patients with Her2 positive disease must have received ≥1 line of anti-Her2 based therapy
* At least 1 measurable or evaluable lesion per RECIST 1.1. Screening imaging must be obtained within 6 weeks of signing the informed consent form
* Completion of systemic therapy at least 7 days before leukapheresis

  o Immune checkpoint inhibitor therapy must be completed at least 14 days before leukapheresis
* Lab requirements (hematology):

  * Absolute neutrophil count ≥1.0 K/mcL
  * Hemoglobin ≥9 gm/dL
  * Platelet count ≥75 K/mcL
  * Blood product transfusion or growth factor support cannot occur within 7 days of testing
* Lab requirements (serum chemistry):

  * Bilirubin ≤1.5× upper limit of normal (ULN)
  * Serum alanine aminotransferase and serum aspartate aminotransferase (ALT/AST) level ≤3× ULN
  * Calculated clearance of ≥50 mL/min by Cockcroft-Gault equation
* Negative screen for infectious disease markers, including hepatitis B core antibody, hepatitis B surface antigen, hepatitis C antibody, HIV 1-2 antibody, HTLV antibody and syphilis antibody

  o Note: Patients with a history of hepatitis B virus infection are eligible if the hepatitis B viral load is undetectable. Patients with a history of hepatitis C virus infection who were treated for hepatitis C and cured are eligible if the hepatitis C viral load is undetectable
* Serum pregnancy test with negative result at screening and preconditioning and must be willing to use effective and reliable contraception for at least 12 months after T cell infusion (for female participants of childbearing age)
* Resolution of all acute toxic effects of any previous therapeutic or palliative chemotherapy, radiotherapy, or surgical procedures to grade ≤1 (CTCAE v5.0), except for neuropathy and alopecia

Inclusion Criteria for lymphodepleting chemotherapy/CAR T cell infusion

* Life expectancy of ≥4 months
* ECOG performance status of 0-1
* At least 1 measurable or evaluable lesion per RECIST 1.1. Screening imaging must be obtained within 4 weeks before the date of lymphodepletion
* Completion of systemic therapy at least 14 days before lymphodepleting chemotherapy

  o Immune checkpoint inhibitor therapy must be completed at least 28 days before lymphodepleting chemotherapy
* Lab requirements (hematology):

  * Absolute neutrophil count ≥1.5 K/mcL
  * Hemoglobin ≥8 gm/dL
  * Platelet count ≥75 K/mcL
* Lab requirements (serum chemistry):

  * Bilirubin ≤1.5× upper limit of normal (ULN)
  * Serum alanine aminotransferase and serum aspartate aminotransferase (ALT/AST) level ≤3× ULN
  * Calculated clearance of ≥50 mL/min by Cockcroft-Gault equation
* Serum pregnancy test with negative result within 7 days of planned lymphodepletion date and must be willing to use effective and reliable contraception for at least 12 months after T cell infusion (for female participants of childbearing age)
* Resolution of all acute toxic effects of any previous therapeutic or palliative chemotherapy, radiotherapy, or surgical procedures to grade ≤1 (CTCAE v5.0), except for neuropathy and alopecia

Participant Exclusion Criteria

Exclusion Criteria for Leukapheresis or Lymphodepleting chemotherapy/CAR T cell infusion: Participants are excluded from enrollment if any of the following criteria apply:

* Pregnant or lactating
* HIV, active hepatitis C virus, or active hepatitis B virus infection, as determined by quantitative PCR (patients who have undergone negative testing prior to leukapheresis do not require repeat testing)
* Receiving therapy for concurrent active malignancy

  * Note: Patients receiving treatment for in situ skin malignancies are not excluded.
  * Patients with any malignancy diagnosed >3 years before that is thought to be curatively treated and/or has a low risk of recurrence are eligible. Patients may continue to receive adjuvant therapy at the time of study enrollment (e.g., adjuvant hormonal therapy for curatively treated breast cancer).
* Known hematologic malignancy requiring treatment in the preceding 5 years or a known history of lymphoid malignancy
* Previous receipt of CAR T cell therapy or any other cellular therapy
* Previous mesothelin-directed therapy Any major abdominal surgery (laparotomy with resection of gastrointestinal tract or organ resection) that is completed <28 days before study enrollment. Patients who have undergone diagnostic laparoscopy can be included in the study without regard to timing
* Untreated or active central nervous system (CNS) metastases (progressing or requiring anticonvulsants or corticosteroids for symptomatic control). Patients with a history of treated CNS metastases are eligible if all of the following criteria are met:

  * Radiographic demonstration of improvement upon completion of CNS-directed therapy and no evidence of interim progression between completion of CNS-directed therapy and the screening radiographic study
  * Completion of radiotherapy ≥4 weeks before the screening radiographic study
* Active autoimmune disease that has required systemic treatment within 1 year before leukapheresis (with the use of disease-modifying agents, corticosteroids, or immunosuppressive drugs)

  o Note: Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
* Receiving daily systemic corticosteroids ≥10 mg of prednisone daily or equivalent or receiving immunosuppressive or immunomodulatory treatment
* Any of the following cardiac conditions:

  * New York Heart Association stage III or IV congestive heart failure
  * Myocardial infarction ≤6 months before enrollment
  * History of myocarditis
  * Serious uncontrolled cardiac arrhythmia, unstable angina, or uncontrolled infection
  * Left ventricular ejection fraction ≤40%
* Active interstitial lung disease/pneumonitis or a history of interstitial lung disease/pneumonitis requiring treatment with systemic steroids
* Baseline pulse oximetry <90% on room air at the screening time point
* Known active infection requiring antibiotic treatment 7 days before leukapheresis

  o Note: Treatment can be delayed at the discretion of the treating physician to allow the patient to recover from the infection.
* Any other medical condition, e.g. fever >38.0 degrees C, that, in the opinion of the PI, may interfere with the subject's participation in or compliance with the study
* Receipt of live, attenuated vaccine within 8 weeks before the planned lymphodepleting chemotherapy date
* Deemed to be noncompliant by the study team for administration of a high-risk treatment agent and for close follow-up after treatment as required by the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of treatment-emergent adverse events | 1 year
  The primary objective of this study is to assess the safety of M28z1XXPD1DNR CAR T cells administered through the peritoneal cavity. CTCAE v5.0 will be used to assess the severity of all treatment-emergent toxicities and adverse events, regardless of reporting requirements
Maximum Tolerated Dose of M28z1XXPD1DNR CAR T cells | Up to 1 year
  Determine the maximum tolerated dose of M28z1XXPD1DNR CAR T cells administered through the peritoneal cavity.

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Ku, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org